CLINICAL TRIAL: NCT06484959
Title: The Effect of Horticultural Therapy Applied to Nursing Home Workers on Depression, Anxiety, Stress and Burnout Levels
Brief Title: The Effect of Horticultural Therapy on Mental Health and Burnout Levels of Nursing Home Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Suheyla YARALI, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: suheylayaralı-3
Record Dates: First submitted 2024-06-12; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Horticultural Therapy; Anxiety; Depression; Stress; Caregivers
Keywords: Horticultural therapy; exhausted; Caregivers; Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Horticultural therapy 1st session (Other): What is horticultural therapy?: the scope of horticultural therapy, information will be given in the nursing home conference room. The training will be done with a power point presentation.In terms of the suitability of the caregivers, the training will be carried out by dividing into 3 groups of 10 people. Training will last 40 minutes. This training will be on Monday
  Interventions: Other: Assigned Interventions
- Horticultural therapy 2st session (Other): Horticultural therapy garden design and principles?: Within the scope of horticultural therapy, information will be given in the nursing home conference room. The training will be done with a power point presentation.In terms of the suitability of the caregivers, the training will be carried out by dividing into 3 groups of 10 people. Training will last 40 minutes. This process will take place with the soil sample sent to agricultural engineering.This training will be on Tuesday
  Interventions: Other: Assigned Interventions
- Horticultural therapy 3st session (Other): The relationship between soil, plants and water: information will be provided by the landscape architect involved in the research. The scope of horticultural therapy, information will be given in the nursing home conference room. The training will be done with a power point presentation.In terms of the suitability of the caregivers, the training will be carried out by dividing into 3 groups of 10 people. Training will last 30 minutes.This process will take place with the soil sample sent to agricultural engineering.This training will be on Wednesday
  Interventions: Other: Assigned Interventions
- Horticultural therapy 4st session (Other): Introduction and characteristics of plants: This information will be provided by the landscape architect involved in the research. The scope of horticultural therapy, information will be given in the nursing home conference room. The training will be done with a power point presentation.In terms of the suitability of the caregivers, the training will be carried out by dividing into 3 groups of 10 people. Training will last 30 minutes. This training will be on Thursday
  Interventions: Other: Assigned Interventions
- Horticultural therapy 5st session (Other): Care and watering techniques: This information will be provided by the landscape architect involved in the research. The scope of horticultural therapy, information will be given in the nursing home conference room. The training will be done with a power point presentation.In terms of the suitability of the caregivers, the training will be carried out by dividing into 3 groups of 10 people. Training will last 30 minutes. This training will be on Friday.
  Interventions: Other: Assigned Interventions
- Horticultural therapy 6st session (Other): Survey analysis in gardens: Samples will be taken from the soil, analyzed, soil examination will be made, and the substances to be fertilized will be determined. This process will take place with the soil sample sent to agricultural engineering.This was done when the caregivers were informed.
  Interventions: Other: Assigned Interventions
- Horticultural therapy 7st session (Other): Preparing the area in the garden for planting was done when the caregivers were informed. The garden created with the drawings made within the scope of the work plan was prepared. Soil is prepared for planting by hoeing and fertilizing.
  Interventions: Other: Assigned Interventions
- Horticultural therapy 8st session (Other): Planting seedlings and seeds in gardens: The information about horticultural therapy, the plants were planted by the caregivers. This process has been achieved by implementing the training and information provided by the researchers.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Assigned Interventions

SUMMARY:
The incidence of people with disabilities in need of care services is increasing all over the world. This situation significantly increases the need for nursing homes and caregivers. In many countries, it is seen that "Horticultural Therapy" programs have started to be implemented to improve mental health. In this context, our aim in the project is to determine the effect of the "Horticultural therapy" program applied to nursing home employees in terms of mental health and burnout in nursing home employees. It is thought that the positive effect of this practice on nursing home employees will be able to better maintain their care-oriented practices. It is envisaged that the gardens to be built within the scope of the therapy program can be planned as areas where both caregivers and caregivers can be used, and the application can be integrated into other areas within the scope of public health over time

DETAILED DESCRIPTION:
Caregivers working in a nursing home will be in the experimental group, and caregivers working in a different care center in the same region will be in the control group. A total of 8 sessions of horticultural therapy activities will be explained to the nursing home employees in the experimental group 1 time a week for 2 months. These trainings, which will be given to the people in the experimental group, will be held in the service building in the nursing home building and in the garden (practical) trainings. 4 different groups of 8/9 people will be formed from 30 people in each garden experiment group and the gardens will be allocated to the users. The purpose of these groups is not to make different applications, but to use the area comfortably. These garden users will be given different vegetables, fruits, seasonal flowers, fruit and ornamental tree seedlings and will be asked to design and implement their own gardens. The preliminary preparation of the gardens will be done through the procurement of services within the scope of the project.Horticultural therapy training will be carried out by the landscape architect who is a researcher in the project. In our project, all activities will be carried out under the supervision of nurse researchers and landscape architect researchers involved in the project. This therapy program is expected to reduce depression, anxiety, stress levels and burnout levels that affect mental health. It is thought that the positive effect of this practice on nursing home employees will be able to better maintain their care-oriented practices. It is envisaged that the gardens to be built within the scope of the therapy program can be planned as areas where both caregivers and caregivers can be used, and the application can be integrated into other areas within the scope of public health over time.

ELIGIBILITY:
Inclusion Criteria:

* Working in a nursing home
* Not being allergic to flowers and plants
* Willingness to work
* To be open to communication and cooperation,
* Scoring 8 points or more on the stress sub-dimension of the DASS measurement tool

Exclusion Criteria:

* Those with musculoskeletal disorders
* Those who use antipsychotic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | [Time Frame: up to 1 day]
  The form consists of 10 questions containing information about caregivers affected by the earthquake created by the researcher within the scope of the literature. The form includes questions including age, gender, education, marital status, number of children, occupation, duration of work in a nursing home, chronic disease status, medication used continuously, social activity with continuous participation, previous psychiatric / psychological help.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale | [Time Frame: up to 10 week ]
  The four-point Likert type scale developed by Lovibond and Lovibond (1995) consists of 14 depression, 14 anxiety and 14 stress dimensions; In order to provide faster, more effective access to resources and more qualified use of time, the short form of the scale, which consists of seven items, consists of 21 items. It is presented in a four-point Likert form as "Not Suitable at All (0) Somewhat Suitable (1) Generally Suitable (2) Completely Suitable (4)" and shows that as the scores obtained from the scale increase, the symptoms of depression, anxiety and stress increase.
The Maslach Burnout Scale | [Time Frame: up to 10 week ]
  developed by Christina Maslach and Susan Jackson (Maslach et al., 1997) and adapted to Turkish and conducted by Ergin (Ergin, 1992), was created to measure the perceived level of burnout. The 7-point Likert type scale, which consists of a total of 22 items and consists of the options 'Never - A few times a year - Several times a month - Once a month - Once a week - Every day" in its original form, was reduced to five options in the adaptation study made by Ergin (1992) on the grounds that it was not suitable for Turkish culture. These options are listed according to their weight as follows: 1-) Never, 2-) Very rare, 3-) Sometimes, 4-) Most of the time, 5-) Always. The Maslach Burnout scale has three sub-dimensions. These; Emotional exhaustion consisting of nine items, depersonalization consisting of five items, and low sense of personal achievement consisting of eight items are subscales.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yarali S, Cengiz M, Kilic D. The effect of mindfulness-based compassionate living training on post-earthquake trauma, grief process, and self-compassion in earthquake-affected university students: a randomized controlled trial. Psychol Health Med. 2025 Sep 2:1-18. doi: 10.1080/13548506.2025.2552963. Online ahead of print. PMID 40892898